CLINICAL TRIAL: NCT02119923
Title: Effects of Working Memory Training in a Depressed and Anxious Sample
Brief Title: Tackling Depression and Anxiety: A Working Memory Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Ingmar Franken, Professor, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2014-04-08; First posted 2014-04-22 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Major Depression; Anxiety Disorder
Keywords: Depression; Anxiety; Working memory; Rumination; Cognitive training; Executive functioning
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders; Depression; Rumination Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Working memory training (Experimental)
  Interventions: Behavioral: Working memory training
- Placebo training (Placebo Comparator)
  Interventions: Behavioral: Placebo training

INTERVENTIONS:
Behavioral: Working memory training — The WM consisted of two tasks; the Number-letter task (Rogers & Monsell, 1995) and an Updating task. The Number-letter task trains the ability to shift between task relevant stimuli. Participants need to shift between four categories. In the Updating task participants receive a set of three words in which they have to compare the two consecutive words on emotional valence (positive or negative) to train their updating skills. Participants executed the training three times a week during four weeks.
  Arms: Working memory training
Behavioral: Placebo training — Both the WM and the placebo training consisted of two tasks; the Number-letter task (Rogers & Monsell, 1995) and an Updating task. To prevent training WM the placebo training was a simplified version of the Number-letter task in which shifting was not required. In the Updating task the placebo group only had to count the number of positive or negative words. Participants executed the training three times a week during four weeks.
  Arms: Placebo training

SUMMARY:
Anxiety and depression are both associated with impairments in executive functions, including working memory (WM) which is needed to maintain and manipulate goal-relevant information. Due to these WM impairments anxious and depressed individuals have difficulties inhibiting and shifting from irrelevant (negative) information and updating goal relevant information. This study explored whether training WM decreases these impairments and reduces clinical symptoms and rumination. Eighty-four individuals diagnosed with major depression and forty-nine individuals with an anxiety diagnosis executed WM or control tasks three times a week, during four weeks. Before, after training and at a two months follow-up measurement depression and anxiety symptoms, WM capacity and rumination behaviour were assessed. Training WM did only result in a reduction of anxiety symptoms in the depression group. These findings are inconsistent with promising results of individual studies showing training WM result in an enlarged WM capacity and a decrease of psychopathological symptoms. However, our results are in line with recent meta-analyses and reviews which show that WM training do not lead to generalized effects and therefore, doubt the clinical relevance of WM training programs.

ELIGIBILITY:
Inclusion Criteria:

* Major depression diagnosis
* Anxiety disorder diagnosis

Exclusion Criteria:

* Current psychosis
* Current substance dependency

Ages: 16 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory Second Edition (BDI-II) score change between pre and post training and at follow-up measurement (2 months after post measurement) | Pre training (baseline), post training (4 weeks after baseline, training starts 1 day after baseline) and follow-up (2 months after post-test)
  Depression is measured with the BDI-II

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) scores change from pre to post training and to follow up measurement (2 months after post measurement) | Pre training (baseline), post training (4 weeks after baseline, training starts 1 day after baseline) and follow-up (2 months after post-test)
  The STAI measures state, trait and total anxiety

OTHER OUTCOMES:
Ruminative Response Scale (RRS) score change between pre and post training and follow up (two months after post) | Pre training (baseline), post training (4 weeks after baseline, training starts 1 day after baseline) and follow-up (2 months after post-test)
  The RRS measures rumination
Symmetry Span score change between pre and post training and at follow-up measurement (2 months after post measurement) | Pre training (baseline), post training (4 weeks after baseline, training starts 1 day after baseline) and follow-up (2 months after post-test)
  The Symmetry Span measures working memory capacity
Internal shift task score change between pre and post training and at follow-up measurement (2 months after post measurement) | Pre training (baseline), post training (4 weeks after baseline, training starts 1 day after baseline) and follow-up (2 months after post-test)
  The internal shift task measures working memory capacity

CONTACTS AND LOCATIONS:
Overall Officials: Elke Geraerts, PhD, Principal Investigator — Erasmus University Rotterdam; Sabine Wanmaker, MSc, Study Director — Erasmus University Rotterdam
Locations (1):
- Erasmus University Rotterdam, Rotterdam, South Holland, Netherlands